CLINICAL TRIAL: NCT02437669
Title: Intranasal Hydromorphone for the Treatment of Acute Pain in Children: A Pilot Study.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Daniel S Tsze, MD, MPH, Assistant Professor of Pediatrics at CUMC, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAP5709
Record Dates: First submitted 2015-05-05; First posted 2015-05-07 (Estimated); Results first posted 2019-05-08 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Pain
Keywords: Intranasal; Hydromorphone; Pediatric; Emergency department
MeSH Terms: conditions — Pain; Emergencies | interventions — Hydromorphone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intranasal hydromorphone (Experimental): Hydromorphone, intranasal. 2 mg/mL concentration. Initial dose: 0.03 mg/kg, maximum single dose 4 mg. Rescue dose: 0.015 mg/kg, maximum single dose 2 mg.
  Interventions: Drug: Hydromorphone

INTERVENTIONS:
Drug: Hydromorphone — To be administered by intranasal route using mucosal atomization device.
  Other Names: Dilaudid

SUMMARY:
Intranasal hydromorphone has been shown to be effective in reducing acute pain in adults. It has not been previously studied in children, but may be a viable option for effectively and safely reducing pain in children by administering an analgesic by the intranasal route.

This study will be a prospective, open-label pilot study of intranasal hydromorphone in children with moderate to severe acute pain presenting to the pediatric emergency department. The investigators aim to describe the amount of pain reduction associated with intranasal hydromorphone, and to determine the optimal dose of intranasal hydromorphone associated with a clinically meaningful improvement in acute pain.

DETAILED DESCRIPTION:
Primary Aim: Determine the change in pain intensity in children with moderate to severe pain who receive intranasal hydromorphone one hour after administration.

Secondary Aim(s): Describe the incidence of minor and major adverse events associated with intranasal hydromorphone in children with acute pain.

The investigators will assess the patient's pain at baseline (prior to study drug administration), then after study drug administration: 5 minutes, 15 minutes, 30 minutes, 45 minutes, 60 minutes, and then every 30 minutes thereafter until 6 hours; administration of non-protocolized rescue medication administration (i.e. administered after first two rescue doses of IN hydromorphone); or discharge from emergency department (whichever comes first). The pain score at 60 minutes will be the primary outcome.

The investigators will evaluate qualitative improvement in pain intensity at 15- and 30-minutes after study drug administration. If there is no improvement, or worsening of pain intensity, at each assessment, an additional rescue dose rescue dose of intranasal hydromorphone will be administered. After 60 minutes, the treating physician may administer any additional rescue medications at their discretion to treat the child's pain.

The patient will be assessed for minor and major adverse events for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 4 to 17 years old, inclusive
* Moderate to severe pain (i.e. FPS-R or vNRS score of 4 or more)
* Requires parenteral opioid analgesic to treat their pain, as decided by treating physician

Exclusion Criteria:

* Allergy or known contraindication to receiving opioids
* Receipt of any opioid or benzodiazepine within preceding 6 hours
* Presence of intranasal obstruction that cannot be cleared readily
* Cannot speak English or Spanish
* Patient unlikely to be able to complete self-report measures of pain or questionnaires
* Known liver or kidney problems
* Currently critically ill
* Chronic pain condition (e.g. sickle cell disease, fibromyalgia)

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Tsze, MD, MPH, Principal Investigator — Columbia University
Locations (1):
- Morgan Stanley Children's Hospital, New York, New York, United States

REFERENCES:
- [Result] Tsze DS, Pan SS, DePeter KC, Wagh AM, Gordon SL, Dayan PS. Intranasal hydromorphone for treatment of acute pain in children: A pilot study. Am J Emerg Med. 2019 Jun;37(6):1128-1132. doi: 10.1016/j.ajem.2019.03.013. Epub 2019 Mar 13. PMID 30902361

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intranasal Hydromorphone
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Intranasal Hydromorphone: Children who received intranasal hydromorphone
Arm/Group | Intranasal Hydromorphone
Number analyzed (Participants) | 35
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 11 [8 to 14]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 26
  White | 5
  Black | 3
  More than one race | 1
Baseline pain score [Mean (Standard Deviation); unit: units on a scale] — Pain was measured using the Faces Pain Scale - Revised (FPS-R). The FPS-R is a self-reported measure of pain that is administered using a picture of 6 different faces lined up in a row, each face representing an escalating degree of pain intensity. The faces, starting from the left-most face and moving towards the right-most face, are scored 0, 2, 4, 6, 8 and 10. A score of 0 represents no pain, a score of 10 represents "very much pain" (i.e. maximum possible pain). More information about the FPS-R can be found here: https://bit.ly/2VPk8GM
  units on a scale | 7 (0.4)

OUTCOME MEASURES:

1. Primary Outcome: Score on Faces Pain Scale - Revised
Description: Pain was measured using the Faces Pain Scale - Revised (FPS-R). The FPS-R is a self-reported measure of pain that is administered using a picture of 6 different faces lined up in a row, each face representing an escalating degree of pain intensity. The faces, starting from the left-most face and moving towards the right-most face, are scored 0, 2, 4, 6, 8 and 10. A score of 0 represents no pain, a score of 10 represents "very much pain" (i.e. maximum possible pain). More information about the FPS-R can be found here: https://bit.ly/2VPk8GM
Time Frame: 1 hour
Population: Decrease in pain score one hour after terminal dose of intranasal hydromorphone administered
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intranasal Hydromorphone
Number analyzed (Participants) | 35
units on a scale | 4.7 [3.7 to 5.7]

2. Secondary Outcome: Number of Minor Adverse Events
Description: Lightheadedness, dizziness; confusion; sleepy, drowsy, tiredness; nausea; vomiting; itchiness, warm sensation; dry mouth; bad taste in mouth; rhinitis.
Time Frame: 6 hours
Measure: Number; unit: Minor adverse events
Arm/Group | Intranasal Hydromorphone
Number analyzed (Participants) | 35
Minor adverse events | 39

3. Secondary Outcome: Number of Major Adverse Events
Description: Oxygen desaturation, respiratory depression, hypotension, bradycardia, need for supplemental oxygen, bag-mask ventilation, airway support intervention, administration naloxone.
Time Frame: 6 hours
Measure: Number; unit: Major adverse events
Arm/Group | Intranasal Hydromorphone
Number analyzed (Participants) | 35
Major adverse events | 0

4. Secondary Outcome: Score on Verbal Numeric Rating Scale
Description: Pain was measured using the Verbal Numerical Rating Scale (VNRS). The VNRS is a self-reported measure of pain that is administered verbally by asking a patient to rate their pain on a scale from 0 to 10, with 0 representing no pain, and 10 representing maximum pain. More information about the VNRS in children can be found here: https://bit.ly/2VZ7aWU
Time Frame: 1 hour
Population: Decrease in pain score one hour after terminal dose of intranasal hydromorphone administered
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intranasal Hydromorphone
Number analyzed (Participants) | 35
units on a scale | 5.1 [4.2 to 6]

ADVERSE EVENTS:
Time Frame: 6 hours
Arm/Group | Intranasal Hydromorphone
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 22/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intranasal Hydromorphone (N=35)
Sleepy, drowsy, or tired (General disorders) | 11
Bad taste in mouth (General disorders) | 8
Lightheaded, dizzy (General disorders) | 8
Dry mouth (General disorders) | 5
Rhinitis (General disorders) | 3
Nausea (General disorders) | 2
Confusion (Nervous system disorders) | 1
Itchiness (Skin and subcutaneous tissue disorders) | 1
Vomiting (Gastrointestinal disorders) | 0
Warm sensation (General disorders) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-16): https://cdn.clinicaltrials.gov/large-docs/69/NCT02437669/Prot_SAP_000.pdf